CLINICAL TRIAL: NCT04836221
Title: Multi-level Interventions to Manage Co-morbidities Among Black Breast and Prostate Cancer Patients
Brief Title: Comorbidities And Reducing inEquitieS
Acronym: CARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Pfizer (Industry); American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Hannah Arem, Scientific Director, Implementation Science, Medstar Health Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 00003543
Record Dates: First submitted 2021-03-24; First posted 2021-04-08 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Cancer, Breast; Diabetes Mellitus; Hypertension; Cancer Prostate
Keywords: Prostate Cancer; Breast Cancer; Diabetes Mellitus; Hypertension; Community Health Workers; mHealth
MeSH Terms: conditions — Breast Neoplasms; Diabetes Mellitus; Hypertension; Prostatic Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Will receive mHealth support for comorbidity and support from a Community Health Worker by phone
  Interventions: Behavioral: Support

INTERVENTIONS:
Behavioral: Support — Community Health Workers will conduct weekly phone calls to monitor blood pressure or blood glucose, to check in on patient need for social, practical or emotional supports, and to encourage healthy lifestyle modification.
  Participants will also have access to a mobile app to support chronic disease management (Either diabetes or hypertension).

SUMMARY:
Black cancer patients tend to have worse outcomes than White cancer patients. Some of this disparity may be due to comorbidities. The purpose of this study is to improve management of co-morbidities among cancer patients in order to improve cancer outcomes and improve health equity.

Comorbidities such as diabetes and hypertension can complicate cancer treatment or can make it difficult to reach optimal health after treatment. This study will offer additional support and tools to manage cancer patient's health needs. First, the study will use a mobile health application, managed by a company called Welldoc, to monitor patient progress in real time and to provide ongoing guidance. Second, the study will connect patients with a Community Health Worker who will speak with them weekly to discuss self-care information, including medical scheduling or appointment needs, and assist with daily self-monitoring of blood pressure and/or blood glucose monitoring. Lastly, an oncology nurse will monitor reported health and triage any medical needs and whether additional medical care is needed.

ELIGIBILITY:
Inclusion Criteria:

* Black women with a diagnosis of stage 0-IV breast cancer and within a month of treatment initiation or with 6+ months of treatment left OR Black men with a history of prostate cancer who are on long-term androgen deprivation therapy;
* Blood pressure >=120/80 OR diagnosis of diabetes
* Individuals who develop these conditions during treatment such as those scheduled to initiate steroid-containing chemotherapy or targeted PI3K inhibitor therapies
* Access to a smartphone and/or internet for the duration of the study.
* Can understand and communicate in English

Exclusion Criteria:

- Unwilling to participate in a 6-month study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of study protocol | Study recruitment period will be approximately 12 months
  Accrual of >50 patients into the study
Feasibility of an active management strategy for comorbidities | Study duration will be 6 months for prostate cancer patients and duration of treatment plus one month for breast cancer patients (approximately 7 months)
  >80% recording blood pressure and/or blood glucose 3+ times per week
Feasibility of an active management strategy for comorbidities | Study duration will be 6 months for prostate cancer patients and duration of treatment plus one month for breast cancer patients (approximately 7 months)
  >80% completion of weekly phone calls with community health workers

SECONDARY OUTCOMES:
Provider perspectives on acceptability of active management of comorbidities | Beginning and end of study (approximately 18 months)
  >80% reporting agree to completely agree on the scale: Acceptability of Intervention Measure (FIM) measure.

OTHER OUTCOMES:
Preliminary changes in self-efficacy | To be assess at baseline and end of study; approximately 6-7 months per participant
  PROMIS Self-Efficacy for Managing Chronic Conditions
Preliminary changes in social support | To be assess at baseline and end of study; approximately 6-7 months per participant
  PROMIS Social Support

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Arem, PhD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States